CLINICAL TRIAL: NCT06068907
Title: Validity and Reliability of Pressure Pain Threshold Assessment in Patients With Elbow Pain
Brief Title: Pain Pressure Threshold in Elbow Pain
Status: Enrolling by invitation | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 333333
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-07

CONDITIONS: Pain, Chronic; Elbow Disease
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Although validity and reliability studies have been completed in different patient groups in the literature, the validity and reliability of pressure pain threshold assessment in patients with elbow pain has not been studied. This study aims to study the validity and reliability of pressure pain threshold assessment in patients with elbow pain.

DETAILED DESCRIPTION:
Unidimensional and multidimensional scales based on patient reporting are mostly used in pain assessment. Although determining pain severity based on patient reporting is important, the patient's physiological and psychological characteristics may make it difficult to interpret the responses. Therefore, objective measurement of pain is very valuable in assessing health status. Another approach to assessing variation in pain perception is to define pressure pain threshold. Although validity and reliability studies have been completed in different patient groups in the literature, the validity and reliability of pressure pain threshold assessment in patients with elbow pain has not been studied. This study aims to study the validity and reliability of pressure pain threshold assessment in patients with elbow pain.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65 years
* Having non-specific elbow joint pain that has been ongoing for the last 3 months
* Having the ability to read and write Turkish
* No vision or hearing problems
* Must have a level of cooperation that can comply with the evaluation

Exclusion Criteria:

* Participated in a physiotherapy program due to elbow problem in the last 6 months
* Presence of neurological or cognitive impairment
* Fractures related to malignant conditions and/or elbow fractures
* Nerve injury, heterotopic ossification or myositis ossificans
* Having elbow arthrosis and/or elbow joint contracture
* Nonunion, malunion and infection problems
* Having complex regional pain syndrome
* Having any known rheumatological, cardiovascular, respiratory or psychiatric disease
* Having a skin disease that will affect the upper extremity evaluation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with elbow pain who volunteer to participate in the study and meet the inclusion criteria will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2025-02-18 (Estimated)

PRIMARY OUTCOMES:
Pressure Pain Threshold | Baseline (First assessment)
  A digital algometer (Commander Algometer, JTECH Medical, USA) will be used. A pressure will be applied to the pulp of the thumb of the hand, which is the control point for the patient to separate the sensation of pain and pressure. Then, a force will be applied to the same point, causing pain. In the supine position, the pressure will be applied vertically to the lateral and medial epicondyle of the humerus, olecranon fossa, radial head, lateral and medial supracondylar foss, biceps, triceps, brachialis and brachioradialis muscle body, increasing the pressure by 1 kg/cm² every three seconds until the patient feels pain. The patient will be asked to report pain as soon as he or she feels it while applying force (kg/cm²) with the device. This process will be repeated three times and there will be a 60-second break between repetitions. The same evaluation will be carried out by a second independent evaluator on the same day, 10 minutes after the first evaluation.

SECONDARY OUTCOMES:
Pressure Pain Threshold | 3 days after the first assessment (Second assessment)
  A digital algometer (Commander Algometer, JTECH Medical, USA) will be used. A pressure will be applied to the pulp of the thumb of the hand, which is the control point for the patient to separate the sensation of pain and pressure. Then, a force will be applied to the same point, causing pain. In the supine position, the pressure will be applied vertically to the lateral and medial epicondyle of the humerus, olecranon fossa, radial head, lateral and medial supracondylar foss, biceps, triceps, brachialis and brachioradialis muscle body, increasing the pressure by 1 kg/cm² every three seconds until the patient feels pain. The patient will be asked to report pain as soon as he or she feels it while applying force (kg/cm²) with the device. This process will be repeated three times and there will be a 60-second break between repetitions.
Pain Intensity | Baseline
  Pain intensity will be measured using the visual analogue scale (VAS). The participants will be asked to indicate their perceived pain at rest, during activity and at night on the 10 cm line between no pain and terrible pain. The score will be determined by measuring the distance on 10 cm line using a ruler. The minimum and maximum possible scores are 0 and 10, with higher scores indicating greater pain intensity.
Functional Status | Baseline
  The functional status of the patients will be evaluated by The Disabilities of the Arm, Shoulder and Hand (DASH). It comprises 30 core questions and optional additional 8 questions that are scored on a 5-point Likert-type scale (no difficulty-unable). The cumulative DASH score is ranged from 0 to 100, where the higher scores indicate an increased degree of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, PT, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)